CLINICAL TRIAL: NCT04853316
Title: Household Transmission Dynamics and Viral Load Among Asymptomatic SARS-CoV-2 Infected Children
Brief Title: Asymptomatic SARS-CoV-2 Detection in Children
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: REB20-0609
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-08

CONDITIONS: Covid19; SARS-CoV-2
Keywords: COVID19; Household transmission; Pediatrics; Asymptomatic; Public health
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — SARS-CoV-2 Testing will be performed according to local public health and institutional guidelines. For any participants who tested positive for the presence of SARS-CoV-2, an aliquot of the corresponding positive test will be obtained. Viral load quantification will be performed on any specimens obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Exposed (SARS-CoV-2 positive): Participants found positive by SARS-CoV-2 testing.
- Control: Unexposed (SARS-CoV-2 negative): Participants found negative by SARS-CoV-2 testing.

SUMMARY:
The primary objective of this study is quantify the transmission risk posted by SARS-CoV-2 in pre/asymptomatic infected children in order to inform the public health response to the COVID-19 pandemic.

DETAILED DESCRIPTION:
1. Background & Rationale:

   Background: Transmission from individuals with pre-symptomatic and asymptomatic (hereafter abbreviated as pre/asymptomatic) SARS-CoV-2 infections is the Achilles' heel of COVID-19 pandemic control1. While pediatric SARS-CoV-2 infection is yet to be fully characterized, and generally children are more likely to experience asymptomatic infection or mild disease compared with adults, severe outcomes are possible. Although person-to-person spread is well described in children, as schools have been closed, the transmission risk in that environment remains unknown. More importantly, the contribution of pre/asymptomatic children to overall transmission of SARS-CoV-2 is unclear with most pediatric cases linked to a symptomatic household member. According to China's National Health Commission, 130 (78%) of 166 new infections identified on April 1, 2020 were asymptomatic. In addition, data from an adult long-term care facility in Washington indicates that symptom-based screening failed to identify a significant proportion of COVID-19 cases. Furthermore, based on RT-PCR cycle threshold values, large quantities of viral RNA were detected in pre/asymptomatic residents, suggesting the potential for transmission regardless of symptoms. Asymptomatic pediatric colonization, while reported, is poorly described.

   Rationale: SARS-CoV-2 shedding has been noted to occur in minimally symptomatic and asymptomatic infected persons. Children therefore, who appear to more commonly experience mild and asymptomatic infection, may represent a significant risk of household and community transmission. Recommendations for school closures are currently based on assumptions as well as evidence gathered from influenza outbreaks where these measures are known to reduce social contacts and interrupt transmission. School closures, however, disrupt the lives of students and their families and may have negative consequences on child health16. Moreover, COVID-19 transmission modelling studies predict that school closures alone prevent only 2 - 4% of COVID-19-related deaths in the general population, much less than other physical distancing interventions. It should be noted that as school closures were in place before observational studies could begin, the secondary clinical attack rate of pre/asymptomatic children is unknown.
2. Research Questions & Objectives:

   The primary objective of this study is quantify the transmission risk posted by SARS-CoV-2 in pre/asymptomatic infected children in order to inform the public health response to the COVID-19 pandemic by determining the following:

   If the proportion of household members who develop symptomatic illness over the subsequent 12 days is greater among households of pre/asymptomatic SARS-CoV-2 positive children relative to negative children. Mathematical models will be developed to understand the risks associated with other community transmission settings.

   In SARS-CoV-2 positive children, if quantitative viral loads differ between those who become symptomatic relative to those who remain asymptomatic and have secondary household cases.

   Secondary aims of this study include the following:

   Determining risk factors for SARS-CoV-2 pre/asymptomatic infection in children.
3. Study Design and Methods:

A prospective cohort study, taking place at multiple institutions throughout the United States and Canada, of children brought to the Emergency Department for care due to a condition or illness unrelated to SARS-CoV-2 infection who are tested as part of ongoing local asymptomatic surveillance programs.

For every SARS-CoV-2-positive asymptomatic child enrolled, three asymptomatic SARS-CoV-2-test negative children will also be recruited.

Any child that is tested for the presence of SARS-CoV-2 who is asymptomatic as part of clinical care, will be potentially eligible for the study. Locally, any child who is tested for the presence of SARS-CoV-2 and who is not displaying any known COVID-19 symptoms will be asked by an Alberta Health Services ED staff member for consent to provide their information to the research team to be contacted about potential participation in the study (consent to contact). Due to testing result timelines and to minimize possible exposure, informed consent/assent will be obtained via telephone and a copy of the consent documentation will be sent via email to the consenting individual, if required. Eligibility for the study based on inclusion and exclusion criteria will be determined over the telephone. Data will be obtained from the participant, their caregiver, and their medical chart, as appropriate. To obtain data related to symptomology, additional medical care, additional testing, and household transmission, a follow up questionnaire will be performed 14 days after the baseline ED visit. If a member of the household is waiting on SARS-CoV-2 testing results at the 14 day follow up time point, an additional call will be made 21 days after the baseline ED visit to obtain SARS-CoV-2 test results. A follow-up call will be performed at 90 days to identify any chronic symptoms that may have developed.

ELIGIBILITY:
Inclusion Criteria:

* Younger than 18 years of age
* Had SARS-CoV-2 NAT testing performed during the ED visit as part of an ongoing active asymptomatic surveillance program:

  1. Exposed (SARS-CoV-2 positive) specific: Was found positive by SARS-CoV-2 NAT testing in the ongoing active surveillance program
  2. Unexposed (SARS-CoV-2 negative/control) specific: Was found negative by SARS-CoV-2 NAT testing in the ongoing active surveillance program

Exclusion Criteria:

* Presence of any of the following viral symptoms commonly associated with SARS-CoV- 2 infection: fever, cough, dyspnea/difficulty breathing, generalized fatigue/weakness, myalgia (muscle or body aches), chills, feeling very unwell, sore throat, runny nose, gastrointestinal symptoms (vomiting, diarrhea), conjunctivitis, headache, anosmia (loss of smell), ageusia (loss of taste) or rash in the 24 hours preceding the index visit (when the child was tested for the presence of SARS-CoV-2).
* Previously diagnosed with SARS-CoV-2 infection based on a positive swab or serology (blood) test.
* Decline to provide informed consent and/or assent, as required

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children younger than 18 years of age presenting to a participating ED who meet institutional surveillance screening guidelines (i.e. present with a non-infectious, non-viral concern) and undergo SARS-CoV-2 testing. The number of children eligible may vary based on evolving SARS-CoV-2 testing procedures, public health policy, and patient volumes.
Sampling Method: Non-Probability Sample
Enrollment: 372 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Symptoms of COVID-19 in household members of participating children in the subsequent 14 days following enrollment | 14 days
  The clinical secondary attack rate (SAR) for households of participating children, which will be compared to generate the relative SAR for households of children with varying case and symptom statuses.

SECONDARY OUTCOMES:
Viral Load of SARS-CoV-2 in positive children | 14 days
  The difference in typical viral loads between children of different symptom and case statuses, as well as those with and without clinical secondary cases.

OTHER OUTCOMES:
Presence of epidemiological risk factors for SARS-CoV-2 infection | 14 days
  Risk factors such as exposures, travel, following public health policy. The frequency of such risk factors among participating children will allow for calculation of the relative risk of such factors.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Freedman, MD, Principal Investigator — University of Calgary
Locations (5):
- United States (4):
  - Children's of Alabama, Birmingham, Alabama
  - University of California, San Diego - Rady Children's Hospital, San Diego, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Medical Center of Dallas - UT Southwestern, Dallas, Texas
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No